CLINICAL TRIAL: NCT05045495
Title: Adult Pilot Study to Establish the Reference Ranges and Optimal Cut-offs for Oral 50g Sucrose Challenge Test & 13C-Sucrose Breath Test for CSID Cases (Previously Diagnosed Sucraid Responders) & Controls (GI Asymptomatic Healthy Volunteers)
Brief Title: Adult Pilot Study for Reference Ranges and Optimal Cut-offs for the Sucrose Challenge Test and Sucrose Breath Test
Status: Completed | Type: Observational
Sponsor: QOL Medical, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SSDXA-12
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Congenital Sucrase-Isomaltase Deficiency
Keywords: CSID
MeSH Terms: conditions — Sucrase-isomaltase deficiency, congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cheek cell samples via buccal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer: 120 Healthy Volunteers will perform the 50-gram sucrose challenge test, Sucrose hydrogen methane breath test, 13C-sucrose breath test and collect buccal swab samples for genetic testing.
  Interventions: Diagnostic Test: Sucrose Hydrogen Methane Breath Test
- CSID Case: 50 CSID cases defined by being on Sucraid for at least 12 months will perform the 50-gram sucrose challenge test, Sucrose hydrogen methane breath test, 13C-sucrose breath test and collect buccal swab samples for genetic testing.
  Interventions: Diagnostic Test: Sucrose Hydrogen Methane Breath Test

INTERVENTIONS:
Diagnostic Test: Sucrose Hydrogen Methane Breath Test — Subjects will collect 2 buccal swabs for the sucrase genetic test and then subjects will simultaneously conduct the sucrose challenge test, sucrose hydrogen methane breath test, and the 13C-sucrose following ingestion of 50-grams of sucrose (table sugar) mixed with 8 ounce of water.
  Other Names: 13C-Sucrose Breath Test; Sucrase Genetic Test (Buccal Swab); Sucrose Challenge Test

SUMMARY:
An adult pilot study to establish the normal reference range and optimal cutoffs for the oral 50g Sucrose Challenge Test (SCT) and the 50g 13C-Sucrose Breath Test (CBT) for patients with CSID and healthy controls. This study will enroll 120 healthy controls and 50 CSID patients. No study drug will be administered during this study.

DETAILED DESCRIPTION:
In an effort to mimic the real-world diagnostic setting for these tests, this study will be conducted virtually using a central site with telemedicine capabilities and electronic data capture software to collect data in real time via a mobile app. Subject will complete 3 visits within 21 days. Eligible subjects will undergo the following tests:

1. 50g 13C-Sucrose Breath Test (CBT)
2. Sucrose Intolerance Hydrogen Methane Breath Test (HBT)
3. Sucrose Challenge Test (SCT)
4. Buccal swab for CSID Genetic Testing (GT)

The primary aim is to establish the reference/normal ranges and optimal cutoff values for the SCT and CBT.

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide informed consent prior to any study procedures being performed.
* Subject is a U.S. resident, and speaks and understands English
* Subject is male or female, ≥ 18 years old.
* CSID Cases must have been on Sucraid for at the last 12 months.
* Healthy Volunteers do not have a CSID diagnosis or other chronic gastrointestinal conditions.
* Subject must have their own Android or Apple device to access the mobile patient app.

Exclusion Criteria:

* Females who are lactating or pregnant.
* Subjects with allergy to sucrose.
* Subjects with causes of abdominal pain or altered bowel habits other than symptoms -related to CSID (in CSID group) such as SIBO, IBD, celiac disease, pancreatitis, or -gastrointestinal bleeding.
* Diabetes mellitus.
* Use of systemic antibiotics, had a barium study, colonoscopy, unexplained runny diarrhea, or similar within 14 days prior to informed consent. Potential subjects can be re-screened once they meet this criterion.
* Recent febrile illness.
* Subject has major physical or psychiatric illness within the last 6 months that in the opinion of the investigator would affect the subject's ability to complete the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and subjects with CSID.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Establish the normal reference range for the 50g Sucrose Challenge Test (SCT) | 4 hours post ingestion of sucrose
  Reference ranges will be estimated by the lower 2.5th percentile and upper 97.5th percentile of the distribution of test results for the case and control populations.
Establish the optimal cutoff values for the 50g Sucrose Challenge Test (SCT) | 4 hours post ingestion of sucrose
  The mean and peak symptom severity score following sucrose ingestion will serve as markers of sucrase activity. The cutoff for the SCT will be determined by the maximum Youden Index that differentiates cases and controls.
Establish the normal reference range for the 50g 13C-Sucrose Breath Test (CBT) | 4 hours post ingestion of sucrose
  Reference ranges will be estimated by the lower 2.5th percentile and upper 97.5th percentile of the distribution of test results for the case and control populations.
Establish the optimal cutoff values for the 50g 13C-Sucrose Breath Test (CBT) | 4 hours post ingestion of sucrose
  The mean and peak symptom severity score following sucrose ingestion will serve as markers of sucrase activity. The cutoff for the SCT will be determined by the maximum Youden Index that differentiates cases and controls.

SECONDARY OUTCOMES:
Compare the positive predictive values (PPV) of the Sucrose Challenge Test (SCT) with the PPV of the Sucrose Hydrogen Methane Breath Test (HBT) | 4 hours post ingestion of sucrose
  PPV of SCT relative to the HBT and percentage of Sucraid® Responders in CSID cases and asymptomatic controls, and in cases confirmed by each of the following three diagnostic tools: HBT, CBT, and SCT.
Compare the negative predictive values (NPV) of the Sucrose Challenge Test (SCT) with the NPV of the Sucrose Hydrogen Methane Breath Test (HBT) | 4 hours post ingestion of sucrose
  NPV of SCT relative to the HBT and percentage of Sucraid® Responders in CSID cases and asymptomatic controls, and in cases confirmed by each of the following three diagnostic tools: HBT, CBT, and SCT.
Compare the positive predictive values (PPV) of the 13C-Sucrose Breath Test (CBT) with the positive predictive value of the Sucrose Hydrogen Methane Breath Test (HBT) | 4 hours post ingestion of sucrose
  PPV of the CBT relative to the HBT and percentage of Sucraid® Responders in CSID cases and asymptomatic controls, and in cases confirmed by each of the following three diagnostic tools: HBT, CBT, and SCT.
Compare the negative predictive value (NPV) of the 13C-Sucrose Breath Test (CBT) with the NPV of the Sucrose Hydrogen Methane Breath Test (HBT) | 4 hours post ingestion of sucrose
  NPV of the CBT relative to the HBT and percentage of Sucraid® Responders in CSID cases and asymptomatic controls, and in cases confirmed by each of the following three diagnostic tools: HBT, CBT, and SCT.

CONTACTS AND LOCATIONS:
Overall Officials: Weng Tao, M.D., Ph. D, Principal Investigator — QOL Medical
Locations (1):
- Science 37-Recruiting Nationally, Culver City, California, United States